CLINICAL TRIAL: NCT01467219
Title: Intra-operative Lymph Node Evaluation Using a Hand Held PET Gamma Probe in Endometrial Cancer Surgery - A Pilot Study
Brief Title: Pilot Study Using a PET Gamma Probe to Evaluate Lymph Nodes in Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11-0211-C
Record Dates: First submitted 2011-10-19; First posted 2011-11-08 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Endometrial Cancer
Keywords: early; high risk
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Lymph Node Excision; Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PET Probe (Experimental): Patients will receive an IV injection of approximately 5 MBq/kg body weight of 18F-FDG (Fludeoxyglucose) (up to 550 MBq). Following injection, patients will undergo CT and PET scans. Intraoperatively, a hand held gamma counter will be used to identify "hot" lymph nodes.
  Interventions: Procedure: lymphadenectomy; Procedure: therapeutic conventional therapy; Procedure: Positron Emission Tomography/ Computed Tomography; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: lymphadenectomy — bilateral pelvic and para-aortic lymph node dissection
Procedure: therapeutic conventional therapy — hysterectomy, bilateral salpingo-oophorectomy,bilateral pelvic and para-aortic lymph node dissection +/- omentectomy via laparotomy, laparoscopy or robotic-assisted
Procedure: Positron Emission Tomography/ Computed Tomography — Pre-operative PET/CT scan
Radiation: fludeoxyglucose F 18 — 5 MBq/kg body weight of FDG (up to 550 MBq)

SUMMARY:
The surgical management of high-risk endometrial cancer often involves an extensive operation to remove lymph nodes as sites of possible cancer spread.

18F-FDG PET/CT imaging is increasingly being used to identify sites of cancer spread and recently groups have used an intra-operative gamma probe to better localize metastatic disease. In this pilot study, patients with newly diagnosed early stage, high-risk endometrial cancer undergoing primary surgery will have a pre-operative PET scan and intra-operative localization of metastatic lymph nodes with the use of a gamma probe. A complete lymphadenectomy will follow and ability to detect positive lymph nodes of both PET scan and the intra-operative probe will be calculated.

This study addresses the feasibility of an FDG detection gamma probe in addition to a pre-operative PET/CT for lymphatic mapping in women with clinical early stage high risk endometrial cancer. The study will also evaluate the role of identifying metastatic lymph nodes intraoperatively that would otherwise be clinically negative.

ELIGIBILITY:
Inclusion Criteria:

* Women with adenocarcinoma of the endometrium with one of the following subtypes:

  * Serous
  * Clear Cell
  * Carcinosarcoma (MMMT)
  * High grade endometrioid
* Clinical stage 1 or 2
* Patients who have signed an approved informed consent.
* Patients who will undergo surgery that includes a hysterectomy and/or hysterectomy, bilateral salpingo-oophorectomy, bilateral pelvic and para-aortic lymph node

Exclusion Criteria:

* Patients with previous retroperitoneal surgery
* Patients with previous history of pelvic/abdominal radiation
* Any patient treated with neoadjuvant chemotherapy and/or radiation

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Identification of metastatic disease in endometrial cancer through pre-operative PET assessment in combination with an FDG intra-operative gamma probe. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Bernardini, MD, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (1):
- University Health Network - Princess Margaret Cancer Center, Toronto, Ontario, Canada